CLINICAL TRIAL: NCT07282860
Title: A Randomized, Controlled Crossover Study on the Safety, Efficacy, and Patient Reported Outcome Measures Comparing the PureWick™ System With an Established Comparator Overnight in the Home Setting for Incontinence in Adult Males
Brief Title: An Evaluation of the PureWick™ Male External Catheter Versus an Established Comparator Overnight in the Home Setting for Incontinence in Adult Males
Acronym: PUREST-M
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UCC-25HC015
Record Dates: First submitted 2025-11-24; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence
Keywords: Male External Catheter; Urine Output Management; Nocturia; Nocturnal Enuresis
MeSH Terms: conditions — Urinary Incontinence; Nocturia; Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Sequence 1 (Experimental): PureWick System used first, followed by crossover to UltraFlex
  Interventions: Device: PureWick System; Device: UltraFlex Self-Adhering Male External Catheter
- Treatment Sequence 2 (Experimental): UltraFlex is used first, followed by crossover to PureWick System
  Interventions: Device: PureWick System; Device: UltraFlex Self-Adhering Male External Catheter

INTERVENTIONS:
Device: PureWick System — The PureWick™ System consists of the PureWick™ Urine Collection System used with the PureWick™ Male External Catheter (MEC), which is intended for non-invasive urine output management in male patients. The PureWick™ MEC is a single-use, non-sterile, commercially available device, which is Class I, 510(K) exempt.
Device: UltraFlex Self-Adhering Male External Catheter — UltraFlex™ is a self-adhering male external catheter used for the drainage of urine. The catheter is applied by the patient or caregiver. The self-adhering male external catheter is designed for the management of adult male urinary incontinence.

SUMMARY:
This post-market study will assess the performance of and user satisfaction with the PureWick™ Male External Catheter in a home setting. The study will also observe safety of the study device and collect information from participants about their experience using the device.

DETAILED DESCRIPTION:
Approximately 100 adult men requiring the use of diapers, pads or equivalent at night for urine management will take part in this prospective, open-label, crossover trial. Participants will be 1:1 randomized to a treatment sequence using two devices: the PureWick™ System (PureWick™ Male External Catheter & PureWick™ Urine Collection System) and the UltraFlex™ Self-Adhering Male External Catheter. Participants will use each urine management device overnight while sleeping for a period of 7 days with a 2-day washout period in between. Total duration of participation is approximately 16 days. The primary endpoint is the mean urine capture rate. The secondary endpoints include the number of device-related AEs requiring medical intervention (safety), device satisfaction and preference questionnaires, and sleep disturbance (quality of life). Capture rates and adverse events are assessed daily throughout each 7-day treatment phase. Patient satisfaction is assessed at the end of each treatment phase. Patient preference is evaluated at study completion. Sleep disturbance is assessed at baseline and every 7 days during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male participants ≥ 18 years of age at the time of signing the informed consent
2. Male anatomy at the time of enrollment
3. Currently use diapers, pads, or equivalent at night for urine output management
4. Willing to comply with all study procedures in this protocol
5. Provision of signed and dated informed consent form

Exclusion Criteria:

1. Has frequent episodes of bowel incontinence; or
2. Has chronic urinogenital infections, active genital herpes; or
3. Has Urinary retention; or
4. Is expected to have an overnight urine output exceeding 1500 mL. This may include, but is not limited to, individuals with polyuria or those receiving diuretic therapy; or
5. Has experience using study devices in the home setting within the last year; or
6. Is agitated, combative, and/or uncooperative and may remove the external catheter; or
7. Has any wound, open lesion or irritation on the genitalia, perineum, or sacrum; or
8. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study; or
9. Is considered a vulnerable population.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Capture rate following void (captured as % of urine captured by device and collected in canister, measured by weight). | From enrollment up to 14 days of treatment
  Prior to each nightly use, the weight of the empty urine collection canister and the weight of a dry absorbent pad are collected. Participants use the device overnight while sleeping with the absorbent pad underneath them. The next morning, the post-void weight of the urine collection canister and the post-void weight of the absorbent pad are collected.
  Capture rate is calculated as the weight of captured urine (post-void canister weight - pre-void canister weight) / total urine volume (captured urine (post-void canister weight - pre-void canister weight) + leaked urine (post-void pad weight - pre-void pad weight)) * 100.

SECONDARY OUTCOMES:
Number of device-related adverse events requiring medical intervention | From enrollment up to 14 days of treatment
  Number of device-related Adverse events requiring medical intervention, such as new prescription medication, surgery or procedure, or therapy ordered by a medical provider to treat or manage the adverse event, in each treatment group.
Participant Device Satisfaction | Day 7 and Day 14, or at the time of treatment discontinuation, whichever comes first.
  Participant experience questionnaire administered after completion of each treatment phase to assess participant device satisfaction. Questions will be scored on a 3-point or 5-point Likert scale with higher scores indicating a better outcome.
Participant Device Preference | Day 15, or at the time of study discontinuation, whichever comes first.
  Participant preference questionnaire administered after completion of both treatment phases to assess preference for the PureWick MEC or UltraFlex sheath-style male external catheter.
Participant Sleep Quality | Starting at baseline and then after Day 7 and after Day 14
  The PROMIS Sleep Disturbance Short Form 4a score collected at baseline and after each 7-day treatment phase. The PROMIS Sleep Disturbance 4a contains 4 scored items each scored from 1 to 5. All item raw scores are computed into a total score where higher scores indicate a worse outcome.

OTHER OUTCOMES:
Device Adherence/Dislodgement | From enrollment up to 14 days of treatment
  Proportion of device wear nights that each device became dislodged.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wagg, Principal Investigator — University of Alberta
Locations (8):
- United States (8):
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - American Institute of Research, Los Angeles, California
  - Finlay Medical Research, Greenacres City, Florida
  - Finlay Medical Research, Miami, Florida
  - Trialfinity Clinical Research Center, Hamilton, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Prime Global Research, The Bronx, New York
  - Monroe Biomedical Research, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No